CLINICAL TRIAL: NCT04335188
Title: COVID-19 Registry Rhineland-Palatinate (Germany) - COVID-19 Disease Registry a National, Multicentre, Non-interventional, Prospective Observational Study
Brief Title: COVID-19 Registry Rhineland-Palatinate (Germany)
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Collaborators: Ministerium für Soziales, Arbeit, Gesundheit und Demografie des Landes Rheinland-Pfalz (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVID-19 Registry
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-patients with SARS-CoV-2 infection: In-patients fulfilling the following criteria:
  SARS-CoV-2 infection In-patient treatment Written informed consent for participation in observational study No explicit medical exclusion criteria are stated to avoid selection bias.
  Interventions: Other: Prospective oberservational registry

INTERVENTIONS:
Other: Prospective oberservational registry — Non interventional study.

SUMMARY:
Documentation of all patients undergoing inpatient treatment for SARS-CoV-2 infection with regard to clinical status at admission, medical history, inpatient treatment and course of disease. The aim is to create a risk stratification of the infection on the basis of clinical data as well as therapy and disease progression of the patients. This may also contribute to a better planning of resources.

ELIGIBILITY:
Inclusion Criteria:

* In-patients fulfilling the following criteria:

SARS-CoV-2 infection In-patient treatment Written informed consent for participation in observational study

Exclusion Criteria:

* No explicit medical exclusion criteria are stated to avoid selection bias.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: About 110 hospitals in Rhineland-Palatinate (Germany) treating patients with SARS-CoV-2 infection.
  All stationary treated patients with SARS-CoV-2 infection will be included.
  Preferably all hospitals in Rhineland-Palatinate, Germany, treating patients with SARS-CoV-2 infection.
  Consecutive enrolment of all patients fulfilling the patient selection criteria to avoid selection bias.
Sampling Method: Non-Probability Sample
Enrollment: 2589 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Chest x-ray | throughout study completion, in average 1.5 years
  presence of infiltrates
Chest CT | throughout study completion, in average 1.5 years
  presence of infiltrates
Supportive care - ICU | throughout study completion, in average 1.5 years
  number of patients with ICU treatment required
Supportive care - oxygen therapy | throughout study completion, in average 1.5 years
  number of patients with oxygen therapy required
Supportive care - ventilation | throughout study completion, in average 1.5 years
  number of patients with ventilation required
Medication | throughout study completion, in average 1.5 years
  number of patients with medication changes
Therapeutic strategies | throughout study completion, in average 1.5 years
  number of patients with ECMO required
Lab parameters | throughout study completion, in average 1.5 years
  number of patients with significant changes in lab parameters
Intra-hospital complications | throughout study completion, in average 1.5 years
  number of patients with complications during hospital stay
Vital status at discharge | throughout study completion, in average 1.5 years
  vital status at discharge: alive, dead

CONTACTS AND LOCATIONS:
Overall Officials: Anselm Gitt, MD, Study Chair — Stiftung IHF and Klinikum der Stadt Ludwigshafen
Locations (1):
- Klinikum der Stadt Ludwigshafen am Rhein GmbH, Klinik für Herzchirurgie, Ludwigshafen, RLP, Germany